CLINICAL TRIAL: NCT06725680
Title: Retrolaminar Block Versus Erector Spinae Plane Block as Opioid-Free Anesthesia for Enhanced Recovery After Posterior Lumbar Discectomy: A Randomized Trial
Brief Title: Retrolaminar Block Versus Erector Spinae Plane Block as Opioid-Free Anesthesia for Enhanced Recovery After Posterior Lumbar Discectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR936/11/24
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Retrolaminar Block; Erector Spinae Plane Block; Opioid-Free Anesthesia; Enhanced Recovery; Lumbar Discectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrolaminar block group (Experimental): Patients will receive retrolaminar block after the induction of general anesthesia.
  Interventions: Other: Retrolaminar block
- Erector spinae plane block group (Experimental): Patients will receive erector spinae plane block after the induction of general anesthesia.
  Interventions: Other: Erector spinae plane block

INTERVENTIONS:
Other: Retrolaminar block — Patients will receive retrolaminar block after the induction of general anesthesia.
  Arms: Retrolaminar block group
Other: Erector spinae plane block — Patients will receive erector spinae plane block after the induction of general anesthesia.
  Arms: Erector spinae plane block group

SUMMARY:
The aim of this study is to compare retrolaminar block and erector spine plane block as opioid-free anesthesia for enhanced recovery after posterior lumbar discectomy.

DETAILED DESCRIPTION:
Lumbar discectomy is a common procedure for patients who experience leg and back pain due to disc problems. Effective pain management is crucial for timely discharge and successful rehabilitation.

Opioid-free anesthesia is a technique that avoids the use of opioids during surgery. Enhanced recovery after surgery (ERAS) pathways are helpful strategies for incorporating opioid-free pain management techniques into clinical practice.

Erector spine plane block (ESPB) and retrolaminar block (RLB) are considered to be compartment blocks or interfacial plane blocks. In these approaches, local anesthetics are assumed to penetrate the superior costotransverse ligament and reach the paravertebral space, although the needle tip is not advanced into the paravertebral space.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Undergoing elective posterior lumbar discectomy under general anesthesia.

Exclusion Criteria:

* Body mass index (BMI) >35 kg/m2.
* Patients with disturbed mental status.
* Allergies to the drugs used in the study.
* Local infection at the puncture site.
* Cardiac insufficiency.
* Renal insufficiency.
* Coagulopathy.
* Chronic opioid use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time from end of surgery to first dose of morphine administrated.

SECONDARY OUTCOMES:
Recovery time | Till first response to verbal command (Up to 1 hour)
  Time from isoflurane discontinuation to the first response to verbal command
Time to discharge | Till the Aldrete score is ≥9 (Up to 3 hours)
  Time from admission to the post-anesthesia care unit (PACU) to discharge from the PACU when the Aldrete score is ≥9) will be recorded.
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4. NRS will be assessed at 0, 4, 6, 8, 12, 18, and 24 h postoperatively.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").
Length of hospital stay | Till discharge from hospital (Up to 1 week)
  Length of hospital stay will be recorded from the admission till discharge from hospital.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication related to the block such as pleural perforation, hematoma, and intraspinal diffusion will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.